CLINICAL TRIAL: NCT06882148
Title: Evaluation of Drug Survival of Target Therapies in Atopic Dermatitis
Brief Title: Drug Survival of Target Therapies in Atopic Dermatitis
Acronym: VADRUDA
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5909
Record Dates: First submitted 2023-10-10; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: target therapies (biological drug, small molecules) — describe the drug sruvival rate of the different approved drugs
  Other Names: selective drugs

SUMMARY:
This is an observational study with drug to evaluate the drug survival of approved target therapies in atopic dermatitis. Patients affected by moderate-severe atopic dermatitis who will start therapy with approved target drugs (dupilumab, tralokinumab, upadacitinib, abrocitinib, baricitinib) for AD will be enrolled. Patients already on therapy with these drugs will also be included.

During the baseline and follow up visits, clinical and demographic data will be collected, according to ordinary clinical practice. Current or retrospective disease severity scores will also be collected.

Among the main: Eczema Area and Severity Index (EASI), Investigator's Global Assessment (IGA), Dermatology Life Quality Index (DLQI), Pruritus Numerical Rating Scale (NRS pruritus), Sleep Numerical Rating Scale (NRS sleep), Patient Oriented Eczema Measure (POEM).

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a chronic, inflammatory skin disease with a prevalence of 10% in adults and 20% in children. It is of primary importance to select the best treatment option as as relapses occur quickly after discontinuation.

Drug survival rate reflects efficacy, tolerability, and safety of a drug, influencing disease management and healthcare costs. AD treatment has been revolutionized by new treatments that include monoclonal antibodies (dupilumab, tralokinumab) and JAK inhibitors (abrocitinib, baricitinib, upadacitinib).

This observational study evaluates the 12-month drug survival of these approved treatments in moderate-to-severe atopic dermatitis, assessing their safety. The study also aims to evaluate the relationship between drug survival and clinical, laboratory, and pharmacological factors.

Patients affected by moderate-severe atopic dermatitis who will start therapy with approved target drugs (dupilumab, tralokinumab, upadacitinib, abrocitinib, baricitinib) for AD will be enrolled. Patients already on therapy with these drugs will also be included.

During the baseline and follow up visits, clinical and demographic data will be collected, according to ordinary clinical practice. Current or retrospective disease severity scores will also be collected.

Among the main: Eczema Area and Severity Index (EASI), Investigator's Global Assessment (IGA), Dermatology Life Quality Index (DLQI), Pruritus Numerical Rating Scale (NRS pruritus), Sleep Numerical Rating Scale (NRS sleep), Patient Oriented Eczema Measure (POEM).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosed with moderate-to-severe atopic dermatitis (EASI>24)
* Undergoing therapy (retrospective cohort) or undertaking systemic therapy with a biological drug or small molecules
* (for retrospective data) presence of at least one follow-up visit after the start of treatment for which clinical and demographic data were collected at baseline and follow-up visits.
* Signature of informed consent to the study and to the processing of personal data for the research

Exclusion Criteria:

* Patients under 18 years of age
* Patients who have undergone systemic therapy with a biological drug or small molecules for whom the start date of treatment is not available and/or no clinical-demographic data were collected at baseline and at follow-up visits.
* Absence of informed consent to the study and processing of personal data for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients affected by moderate-severe atopic dermatitis undergoing target therapies for AD (upadacitinib, baricitinib, abrocitinib, dupilumab, tralokinumab)
Sampling Method: Probability Sample
Enrollment: 1167 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
drug survival evaluation | 1 year
  evaluate the 12-month drug survival rate, for each of the 5 biological drugs/small molecules under study.

SECONDARY OUTCOMES:
drug survival related to safety | through study completion, an average of 3 year
  Number of participants with treatment-related adverse events
relationship between drug survival and clinical data | through study completion, an average of 3 year
  Evaluate the relationship between drug survival and clinical, laboratory and pharmacological determinants.

CONTACTS AND LOCATIONS:
Overall Officials: Ketty Peris, Prof, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- fondazione policlinico universitario agostino gemelli IRCCS, Rome, Italy